CLINICAL TRIAL: NCT02173912
Title: Open-label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetics and Safety Following Administration of CJ-30059 and Co-administration of Candesartan Cilexetil and Amlodipine Besylate in Healthy Volunteers.
Brief Title: Bioequivalence Study of CJ-30059
Acronym: CCA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_CCA_102
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — candesartan cilexetil; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Single-dose crossover
  1. Test: CJ-30059
  2. Reference: Candesartan cilexetil 16 mg and Amlodipine besylate 10mg
  Once daily Oral administration with at least 14 days of washout period
  Interventions: Drug: Candesartan cilexetil 16 mg and Amlodipine besylate 10mg (Reference); Drug: CJ-30059 (Test)
- Sequence 2 (Experimental): Single-dose crossover
  1. Reference: Candesartan cilexetil 16 mg and Amlodipine besylate 10mg
  2. Test: CJ-30059
  Once daily Oral administration with at least 14 days of washout period
  Interventions: Drug: Candesartan cilexetil 16 mg and Amlodipine besylate 10mg (Reference); Drug: CJ-30059 (Test)

INTERVENTIONS:
Drug: Candesartan cilexetil 16 mg and Amlodipine besylate 10mg (Reference) — Sequence 1 receives Candesartan cilexetil 16 mg and Amlodipine besylate 10mg first, then CJ-30059 second, with at least 14-day wash-out period in between.
  Sequence 2 receives CJ-30059 first, then Candesartan cilexetil 16 mg and Amlodipine besylate 10mg second, with at least 14-day wash-out period in between.
Drug: CJ-30059 (Test) — Sequence 1 receives Candesartan cilexetil 16 mg and Amlodipine besylate 10mg first, then CJ-30059 second, with at least 14-day wash-out period in between.
  Sequence 2 receives CJ-30059 first, then Candesartan cilexetil 16 mg and Amlodipine besylate 10mg second, with at least 14-day wash-out period in between.

SUMMARY:
This study is designed to evaluate the bioequivalence of the two treatments, the administration of CJ-30059 and the co-administration of candesartan cilexetil and amlodipine besylate, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 19 and 55 years old(inclusive)
* Body mass index (BMI) in the range of 18.5 to 27 kg/m2(inclusive)
* Available for the entire study period
* Understand the requirements of the study and voluntarily consent to participate in the study

Exclusion Criteria:

* Subjects with a history of gastrointestinal diseases which might significantly change absorption, distribution, metabolism and excretion (ADME) of medicines
* Systolic blood pressure outside the range of 100 to 150 mmHg or diastolic blood pressure outside the range of 70 to 1000 mmHg for male subjects during screening
* Subject with symptoms of acute disease within 14days prior to study drug administration
* Subjects with a history of clinically significant allergies
* Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects whose clinical laboratory test values are outside the accepted normal range. Especially, aspartate aminotransferase (AST) or alamin aminotransferase (ALT) >1.5 times of the Upper Normal Limit or total bilirubin > 1.5 times of the Upper Normal Limit)
* History of drug abuse
* History of caffeine, alcohol, smoking abuse

  * caffeine(coffee, tea, coke) or grapefruit juice > 4 cups/day
  * smoking > 20 cigarettes/day
  * alcohol > 140 g/week
* Positive test results for Hepatitis B antibodies, Hepatitis C virus antibody, and Syphilis regain test
* Participation in any clinical investigation within 30 days prior to study drug administration
* Subjects with whole blood donation within 60 days, component blood donation within 30days and blood transfusion within 30 days prior to study drug administration
* Subjects who are judged unsuitable by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Area Under the plasma concentration-time Curve (AUC_last) of Amlodipine | Upto 72 hours
Area Under the plasma concentration-time Curve (AUC_last) of Candesartan | Upto 72 hours
Maximum plasma concentration (Cmax) of Amlodipine | Upto 72 hours
Maximum plasma concentration (Cmax) of Candesartan | Upto 72 hours

SECONDARY OUTCOMES:
Time to maximum plasma concentration of Amlodipine | Upto 72 hours
Time to maximum plasma concentration of Candesartan | Upto 72 hours
Elimination half-lie of Amlodipine | Upto 72 hours
Elimination half-lie of Candesartan | Upto 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jae-wook Ko, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea